CLINICAL TRIAL: NCT00922753
Title: The Efficacy and Tolerability of Different Levels of Inspiratory Support and PEEP During Preoxygenation. A Randomized Controlled Trial.
Brief Title: Inspiratory Support Improves Preoxygenation in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Tanoubi Issam, M.D., Maisonneuve-Rosemont Hospital, Department Of Anesthesiology
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 06109
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Preoxygenation; Inspiratory; Support; Healthy; EndtidalO2
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BiPAP6 assisted preoxygenation (Active Comparator)
  Interventions: Other: AI-6/PEEP-4
- BiPAP4 assisted preoxygenation (Active Comparator)
  Interventions: Other: AI-4/PEEP-4
- Standard preoxygenation (VS) (Active Comparator)
  Interventions: Other: VS

INTERVENTIONS:
Other: VS — Spontaneous breathing of 100% oxygen in a facemask for 3 minutes
  Arms: Standard preoxygenation (VS)
Other: AI-4/PEEP-4 — Spontaneous breathing of 100% oxygen in a facemask with application of an inspiratory pressure of 4 cm H2O and a positive end-expiratory pressure of 4 cm H2O, for 3 minutes
  Arms: BiPAP4 assisted preoxygenation
Other: AI-6/PEEP-4 — Spontaneous breathing of 100% oxygen in a facemask with application of an inspiratory pressure of 6 cm H2O and a positive end-expiratory pressure of 4 cm H2O, for 3 minutes.
  Arms: BiPAP6 assisted preoxygenation

SUMMARY:
Preoxygenation optimizes oxygen content in the functional residual capacity (FRC). Adequate preoxygenation is defined by an expiratory oxygen fraction (FEO2) > 90%. Inspiratory support and positive end expiratory pressure (PEEP) can create a better reservoir, improve gas exchange and shorten the time needed for adequate preoxygenation. The goal of the study is to evaluate the efficacy and tolerability of different levels of inspiratory support and positive end expiratory pressure during preoxygenation in healthy subjects.

DETAILED DESCRIPTION:
We conducted a double blind prospective randomized trial on 20 healthy volunteers. Each subject went through three modes of preoxygenation in random order: normal breathing (SP), breathing under inspiratory support 4 cmH2O/PEEP 4 cmH2O (PSM-4) and inspiratory support 6 cmH2O /PEEP 4 cmH2O (PSM-6). Each mode lasted for 3 min and parameters were recorded every 10 s. We evaluated subject's tolerance, leaks and easiness of each mode of preoxygenation according to a simplified (1 to 4) scale. Two-way ANOVA was used to compare FEO2 while simple ANOVA was used for time to reach FEO2=90%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged between 20 to 40 years

Exclusion Criteria:

* Body mass index > 30
* Mustache, beard
* Claustrophobia

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
expiratory oxygen fraction (end-tidal 02)

SECONDARY OUTCOMES:
inspiratory oxygen fraction
end-tidal CO2
tidal volume
inspiratory pressure
subject's tolerance
leaks around the mask during preoxygenation
minute volume
endexpiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Issam Tanoubi, M.D., Principal Investigator — Maisonneuve Rosemont Hospital, University Of Montreal; François Donati, PhD, MD, FRCPC, Study Director — Maisonneuve Rosemont Hospital, University Of Montreal; Pierre Drolet, MD, FRCPC, Study Chair — Maisonneuve Rosemont Hospital, University Of Montreal; Louis Phillipe Fortier, MSc, MD, FRCPC, Principal Investigator — Maisonneuve Rosemont Hospital, University Of Montreal
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] HAMILTON WK, EASTWOOD DW. A study of denitrogenation with some inhalation anesthetic systems. Anesthesiology. 1955 Nov;16(6):861-7. doi: 10.1097/00000542-195511000-00004. No abstract available. PMID 13268902
- [Background] Goldberg ME, Norris MC, Larijani GE, Marr AT, Seltzer JL. Preoxygenation in the morbidly obese: a comparison of two techniques. Anesth Analg. 1989 Apr;68(4):520-2. No abstract available. PMID 2494907
- [Background] Gagnon C, Fortier LP, Donati F. When a leak is unavoidable, preoxygenation is equally ineffective with vital capacity or tidal volume breathing. Can J Anaesth. 2006 Jan;53(1):86-91. doi: 10.1007/BF03021532. PMID 16371614
- [Background] Bourgain JL. [Preoxygenation and upper airway patency control]. Ann Fr Anesth Reanim. 2003 Aug;22 Suppl 1:41s-52s. doi: 10.1016/s0750-7658(03)00125-4. French. PMID 12943861
- [Background] Valentine SJ, Marjot R, Monk CR. Preoxygenation in the elderly: a comparison of the four-maximal-breath and three-minute techniques. Anesth Analg. 1990 Nov;71(5):516-9. doi: 10.1213/00000539-199011000-00011. PMID 2221412
- [Background] Byrne F, Oduro-Dominah A, Kipling R. The effect of pregnancy on pulmonary nitrogen washout. A study of pre-oxygenation. Anaesthesia. 1987 Feb;42(2):148-50. doi: 10.1111/j.1365-2044.1987.tb02987.x. PMID 3826588
- [Background] Gambee AM, Hertzka RE, Fisher DM. Preoxygenation techniques: comparison of three minutes and four breaths. Anesth Analg. 1987 May;66(5):468-70. No abstract available. PMID 3578856
- [Background] Hirsch J, Fuhrer I, Kuhly P, Schaffartzik W. Preoxygenation: a comparison of three different breathing systems. Br J Anaesth. 2001 Dec;87(6):928-31. doi: 10.1093/bja/87.6.928. PMID 11878698
- [Background] Machlin HA, Myles PS, Berry CB, Butler PJ, Story DA, Heath BJ. End-tidal oxygen measurement compared with patient factor assessment for determining preoxygenation time. Anaesth Intensive Care. 1993 Aug;21(4):409-13. doi: 10.1177/0310057X9302100406. PMID 8214545
- [Background] Russell GN, Smith CL, Snowdon SL, Bryson TH. Pre-oxygenation and the parturient patient. Anaesthesia. 1987 Apr;42(4):346-51. doi: 10.1111/j.1365-2044.1987.tb03972.x. PMID 3592155
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Baraka A, Haroun-Bizri S, Khoury S, Chehab IR. Single vital capacity breath for preoxygenation. Can J Anaesth. 2000 Nov;47(11):1144-6. doi: 10.1007/BF03027970. PMID 11097548
- [Background] Baraka AS, Taha SK, El-Khatib MF, Massouh FM, Jabbour DG, Alameddine MM. Oxygenation using tidal volume breathing after maximal exhalation. Anesth Analg. 2003 Nov;97(5):1533-1535. doi: 10.1213/01.ANE.0000082528.93345.B9. PMID 14570682
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Wax DB. Mechanism of benefit of head-up preoxygenation in obese patients. Anesthesiology. 2006 Feb;104(2):381; author reply 381. doi: 10.1097/00000542-200602000-00035. No abstract available. PMID 16436870
- [Background] Pelosi P, Ravagnan I, Giurati G, Panigada M, Bottino N, Tredici S, Eccher G, Gattinoni L. Positive end-expiratory pressure improves respiratory function in obese but not in normal subjects during anesthesia and paralysis. Anesthesiology. 1999 Nov;91(5):1221-31. doi: 10.1097/00000542-199911000-00011. PMID 10551570
- [Background] Berthoud MC, Peacock JE, Reilly CS. Effectiveness of preoxygenation in morbidly obese patients. Br J Anaesth. 1991 Oct;67(4):464-6. doi: 10.1093/bja/67.4.464. PMID 1931404